CLINICAL TRIAL: NCT03595020
Title: Probing Prefrontal Cortex Hemodynamic Alterations During Facial Emotion Recognition for Major Depression Disorder Through Functional Near-infrared Spectroscopy
Brief Title: Probing Prefrontal Cortex Hemodynamic Alterations for Major Depression Disorder
Acronym: MDD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20172012-1
Record Dates: First submitted 2018-06-24; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-02

CONDITIONS: Depressive Disorder, Major
Keywords: major depression disorder; functional near-infrared spectroscopy; facial emotion recognition
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MDD group: The major depression group (MDD group) received antidepressant treatment but did not interfere with drug selection.
- HC group: The healthy control group (HC group) don't accept intervention and treatment.

SUMMARY:
Major depression disorder (MDD) has high estimated lifetime prevalence rates of 16.6%. Currently, the diagnosis for the MDD mainly depends on patients' reports of symptoms, observed behaviors and disease course. Establishment of clinically useful biomarkers for the MDD diagnosis would enhance patient management and treatment effect, and lead to the therapies adjusted to the individual. However, no such biomarkers have been established up to now. Therefore, the development of objective and feasible biomarkers is of special significance and a great challenge for accurate and early diagnosis and treatment of depression, in order to overcome the limitations of relying on clinical interviews alone.The ability to correctly recognize emotional states from faces is instrumental for interpersonal engagement and social functioning. Impairments processing of facial emotional expressions and biased facial emotion detection are frequently found in the MDD patients. To date, the studies on neural mechanism of the facial emotion recognition of the MDD patients were mainly based on the functional magnetic resonance imaging (fMRI). Functional near-infrared spectroscopy (fNIRS) has not been applied for the facial emotion recognition for the depression patients up to now. To bridge the important gap in the literature, we used the fNIRS methodology to investigate the neural mechanisms of facial emotion recognition for the patients with depression. We hypothesize the physiological feature of the hemodynamic responses in prefrontal cortex measured by fNIRS under the task of face emotion recognition, including the difference of the median, the Mayer wave power, the mean cross wavelet coefficient, and the mean wavelet coherence coefficient, combined with the behavior measurement (behavior accuracy and response time), could provide a reliable and feasible diagnosis approach to differentiate patients with the MDD from healthy control (HC) subjects with acceptable sensitivity and specificity.

DETAILED DESCRIPTION:
The fMRI technique for functional imaging were limited by the fact that the individuals need to be placed in an uncomfortable or unnatural setting and foreign, noisy, dark, or claustrophobic environment (e.g., lying in a supine position in a narrow gantry with the head restrained during the entire examination), for accurate measurement during the procedure, with relatively lower temporal resolution. In contrast, a multi-channel fNIRS machine provides a completely non-invasive, quiet and mobile measurement of brain function in ordinary clinical settings and allows patients to be comfortably seated in a normal posture in a well-lit room, with higher temporal resolution making it possible to obtain a recording of the actual time course of a hemodynamic epoch in response to a specific cognitive task (e.g., facial emotion recognition task in our study) in a single trial. Additionally, due to the small operating and maintenance costs associated with NIRS, it is possible to run fNIRS study with a large sample of participants.

ELIGIBILITY:
Inclusion Criteria:

* MDD group:

All subjects were free of psychotropic medication for a minimum of 4 weeks; Psychiatric diagnosis was determined by DSM-IV criteria; Depressed subjects were included with 17-item Hamilton Rating Scale for Depression (HRSD) scores ≥ 18; Mini-mental State Examination(MMSE) ≥ 24; All subjects had normal or corrected-to-normal vision.

* HC group:

All subjects were free of psychotropic medication for a minimum of 4 weeks; All subjects did not have any mental, neurological or physical diseases；HRSD scores ≤ 7; MMSE ≥ 28; All subjects had normal or corrected-to-normal vision.

Exclusion Criteria:

* Exclusion criteria were any history of neurologic trauma resulting in loss of consciousness, any current neurologic disorder, any lifetime psychiatric disorder other than major depression in the MDD subjects, or any lifetime psychiatric disorder in control subjects. Careful attention was paid to excluding substance abuse disorders.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study was performed in Xijing Hospital and Xi'an Jiaotong University in China. 100 right-handed subjects meeting DSM-IV criteria for major depression were recruited by advertisement to participate in the study, and were matched with a control group of 100 comparison subjects of university staff members, university students and members of the general population.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale-17(HAMD-17) score alterations | Change from baseline HAMD-17 scores at 6 months
  The HAMD-17 scores are to evaluate the severity degree of depression, and the HAMD-17 scores reduction rate is used to evaluate the clinical treatment effect. If the reduction rate exceeds 50%, it indicates that the clinical treatment is effective.

SECONDARY OUTCOMES:
facial emotion recognition | Difference at facial emotion recognition between day 1 and month 6.
  The ability to correctly recognize emotional states from faces is instrumental for interpersonal engagement and social functioning. Impairments processing of facial emotional expressions and biased facial emotion detection are frequently found in the MDD patients. Functional near-infrared spectroscopy (fNIRS) has not been applied for the facial emotion recognition for the depression patients up to now.
Pittsburgh Sleep Quality Index（PSQI） | Difference at PSQI between day 1, month 3 and month 6.
  PSQI was used to assess the quality of sleep for subjects in the recent month. The total score ranges from 0 to 21 points. The higher the score, the worse the sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Huaning Wang, doctorate, Study Chair — Department of psychiatry, Xijing Hospital
Locations (1):
- Department of psychiatry, Xijing Hospital; Research Institute of Biomedical Engineering, Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zwick JC, Wolkenstein L. Facial emotion recognition, theory of mind and the role of facial mimicry in depression. J Affect Disord. 2017 Mar 1;210:90-99. doi: 10.1016/j.jad.2016.12.022. Epub 2016 Dec 19. PMID 28024224
- [Background] Tsuchida A, Fellows LK. Are you upset? Distinct roles for orbitofrontal and lateral prefrontal cortex in detecting and distinguishing facial expressions of emotion. Cereb Cortex. 2012 Dec;22(12):2904-12. doi: 10.1093/cercor/bhr370. Epub 2012 Jan 5. PMID 22223852
- [Background] Takizawa R, Fukuda M, Kawasaki S, Kasai K, Mimura M, Pu S, Noda T, Niwa S, Okazaki Y; Joint Project for Psychiatric Application of Near-Infrared Spectroscopy (JPSY-NIRS) Group. Neuroimaging-aided differential diagnosis of the depressive state. Neuroimage. 2014 Jan 15;85 Pt 1:498-507. doi: 10.1016/j.neuroimage.2013.05.126. Epub 2013 Jun 10. PMID 23764293